CLINICAL TRIAL: NCT06708793
Title: Environmental Exposures and Sudden Unexpected Infant Death : a Descriptive Study From the French Prospective Multisite Registry (OMIN)
Brief Title: Environmental Exposures and Sudden Unexpected Infant Death
Acronym: ExpoMIN
Status: Active, not recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: AXA Assurances VIE Mutuelle (Unknown); ANSES (Other)
Responsible Party: Sponsor
Other Study IDs: RC23_0513
Record Dates: First submitted 2024-11-26; First posted 2024-11-27 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Sudden Unexpected Infant Death, Air Pollution, Pesticides
Keywords: Sudden unexpected infant death; Sudden infant death syndrome; Perinatal death
MeSH Terms: conditions — Sudden Infant Death; Perinatal Death

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project is a descriptive study designed to identify the exposure of infants who died of MIN to ambient air pollutants, and to measure pesticide concentrations in biological matrices (hair, serum, LCS) within a sample from the OMIN registry. French national registry of STUDY of Sudden Unexpected Infant Death.

DETAILED DESCRIPTION:
This project is a descriptive study designed to estimate the exposure of infants who died of MIN to ambient air pollutants, and to measure pesticide concentrations in biological matrices (hair, serum, LCS) within a sample from the OMIN registry. These two types of pollutants represent two important determinants of environmental health. Although their emission sources and chemical composition differ, these pollutants carry the risk of multiple toxicities that can contribute to the occurrence of Unexpected Infant Death Syndrome (SUID), and are widely present in France, in the air as well as in food, waterways, soils, etc. These two approaches have enabled us to develop two complementary methodologies: geostatistics associated with environmental epidemiology for air pollutants, and analytical environmental chemistry for pesticides.

In addition to matching these exposure measurements with data from the OMIN registry, we will be able to address the impact and determinants of these exposures - i.e., to highlight the individual and collective characteristics that favor high exposure, and to address the toxicological mechanisms linked to these exposures and that may contribute to the occurrence of SUID in general.

ELIGIBILITY:
Inclusion Criteria:

* Died and include in French registry of sudden infant death syndrome

Exclusion Criteria:

* None

Min Age: 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The entire population concerns infants who died of MIN and are included in the OMIN registry. For the ambient air pollution axis, the inclusion criterion is the availability of geolocation (GPS) of the residence. For the pesticides axis, the inclusion criterion is the presence of biological samples in the 3 matrices of interest: serum, hair and cerebrospinal fluid.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Modeling cumulative exposure to several contaminants in ambient air, to ambient temperature in France and to pesticides through proximity to crops, and cross-referencing with data from the OMIN registry | one year

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France